CLINICAL TRIAL: NCT04360486
Title: Expanded Access Protocol For The Treatment Of CORONAVIRUS DISEASE 2019 (COVID-19) With Anti-Sars-CoV-2 Convalescent Plasma (ASCoV2CP)
Brief Title: Treatment Of CORONAVIRUS DISEASE 2019 (COVID-19) With Anti-Sars-CoV-2 Convalescent Plasma (ASCoV2CP)
Status: No longer available | Type: Expanded Access
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: S-20-02; IND 19930 (Other: FDA)
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Anti-Sars-CoV-2 Convalescent Plasma — Fresh frozen plasma, Plasma Frozen for 24 hours (PF-24), or Liquid plasma

SUMMARY:
This treatment protocol is designed to provide convalescent plasma as a therapeutic option for patients diagnosed with and hospitalized for COVID-19 with symptoms ranging from mild to life-threatening.

DETAILED DESCRIPTION:
This is an expanded access open-label, single-arm, multi-site protocol to provide convalescent plasma as a treatment for patients diagnosed with and hospitalized for COVID-19 with symptoms ranging from mild to life-threatening. Efficacy of this treatment will not be evaluated. A single site will initially be established. When additional patients needing therapy are identified at other health care facilities, Force Health Protection (FHP) will send a protocol package, and a site will be established and approved by the Headquarters USAMRDC Institutional Review Board (HQ IRB).

ELIGIBILITY:
Inclusion Criteria:

A patient must meet the following criteria to be included in this protocol:

* DoD personnel covered by the Force Health Protection (FHP) program under the Department of Defense Instruction (DoDI) 6200.02 (active duty service members OCONUS and CONUS) and non-DoD personnel who may be treated for COVID-19 at Military Treatment Facilities (MTFs) under the authority of DoDI 6200.03, including Military Health System (MHS) beneficiaries, patients admitted to MTFs, and patients cared for under defense support for civilian authorities (e.g. hospital ships, field hospitals deployed for the COVID-19 response).
* Laboratory confirmed COVID-19 diagnosis

  * Both PCR and antigen tests are considered to be diagnostic
  * Serum antibody titer testing is not considered to be diagnostic, as patients who recently recovered from COVID-19 will still test positive)
* Hospitalized with symptoms ranging from mild to life-threatening
* Informed consent provided by the patient or legally authorized representative (LAR), except in situations described in 21 CFR 50.23
* Understands and agrees to comply with planned protocol procedures

In general, adults with SARS-CoV-2 infection can be grouped into the following severity of illness categories. However, the criteria for each category may overlap or vary across clinical guidelines and clinical trials, and a patient's clinical status may change over time.

* Asymptomatic or Presymptomatic Infection: Individuals who test positive for SARS-CoV-2 using a virologic test (i.e., a nucleic acid amplification test or an antigen test) but who have no symptoms that are consistent with COVID-19.
* Mild Illness: Individuals who have any of the various signs and symptoms of COVID-19 (eg, fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell) but who do not have shortness of breath, dyspnea, or abnormal chest imaging.
* Moderate Illness: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have saturation of oxygen (SpO2) ≥94% on room air at sea level.
* Severe Illness: Individuals who have SpO2 <94% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, respiratory frequency >30 breaths/min, or lung infiltrates >50%.
* Critical Illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction.

Exclusion Criteria:

Patients who have a medical contraindication for plasma transfusion will be excluded from participation in this protocol. Any patient not meeting the inclusion criteria will not be eligible to receive this treatment. Patients will not be excluded because of receipt of another COVID-19 treatment(s) unless the principal investigator (treating physician) feels that the patient would be put at risk by receiving multiple therapies.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (38):
- United States (26):
  - Naval Hospital Camp Pendleton, Oceanside, California
  - Navy Medical Center San Diego, San Diego, California
  - USS Abraham Lincoln, San Diego, California
  - USS Carl Vinson, San Diego, California
  - USS Essex, San Diego, California
  - USS Makin Island, San Diego, California
  - USS Nimitz, San Diego, California
  - USS Theodore Roosevelt, San Diego, California
  - Evans Army Community Hospital, Fort Carson, Colorado
  - Eglin Air Force Base, Eglin Air Force Base, Florida
  - Naval Hospital Jacksonville, Jacksonville, Florida
  - Martin Army Community Hospital, Fort Benning, Georgia
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Keesler Medical Center, Biloxi, Mississippi
  - Nellis Air Force Base, Las Vegas, Nevada
  - Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina
  - Wright Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - William Beaumont Army Medical Center, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Naval Surface Force Atlantic, Norfolk, Virginia
  - USS Dwight D. Eisenhower, Norfolk, Virginia
  - USS Gerald R. Ford, Norfolk, Virginia
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Lakewood, Washington
- Craig Joint Theatre Hospital Bagram AFGH, Bagrām, Afghanistan
- Djibouti Expeditionary Medical Facility, Djibouti, Djibouti
- Landstuhl Regional Medical Center, Landstuhl, Germany
- Naval Hospital Guam, Hagåtña, Guam
- Baghdad Diplomat Support Center Iraq, Baghdad, Iraq
- Japan (6):
  - Misawa Air Force Base, Aomori
  - Yokota Air Base, Fussa
  - US Naval Hospital Okinawa, Okinawa
  - Naval Hospital Yokosuka, Yokosuka
  - USS America, Yokosuka
  - USS Ronald Reagan, Yokosuka
- US Military Hospital Kuwait, Kuwait City, Kuwait